CLINICAL TRIAL: NCT04661553
Title: Mueller Polarimetric Colposcopy for High-performance Detection of Cervical Changes During Pregnancy (COLPOTERME)
Brief Title: Mueller Polarimetric Colposcopy for High-performance Detection of Cervical Changes During Pregnancy
Acronym: COLPOTERME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191010; 2020-A01932-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-10-23; First posted 2020-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related; Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1: patients with a low risk of premature birth (Experimental): Asymptomatic patient receiving usual follow-up in the maternity ward.
  Interventions: Device: Mueller's polarimetric colposcopy "Group 1"
- Group2: patients with a high risk of premature birth (Experimental): Symptomatic patients with cervical changes objectified by endovaginal ultrasound of the cervix with length <20mm. Asymptomatic patients with a history of premature delivery or late miscarriage and cervical changes objectified by endovaginal ultrasound of the cervix with length <20mm.
  Interventions: Device: Mueller's polarimetric colposcopy "Group 2"

INTERVENTIONS:
Device: Mueller's polarimetric colposcopy "Group 1" — Determination of the best "polarimetric biomarkers" reflecting the status of the cervical microstructure throughout its remodeling process due to the pregnancy in a population with a low-risk premature birth. This "polarimetric biomarkers" should make it possible to accurately determine the time remaining before childbirth for a normal pregnancy and, therefore, to monitor the regular advancement of the gestation.
  Arms: Group1: patients with a low risk of premature birth
Device: Mueller's polarimetric colposcopy "Group 2" — Determination of the best "polarimetric biomarkers" reflecting the status of the cervical microstructure throughout its remodeling process due to the pregnancy in a population at high-risk of preterm birth.
  This "polarimetric biomarkers" should make it possible to accurately determine the time remaining before childbirth for an abnormal pregnancy and, therefore, to predict premature childbirth.
  Arms: Group2: patients with a high risk of premature birth

SUMMARY:
Mueller polarimetric colposcopy appears to be a powerful tool for evaluating cervical microstructure modification during pregnancy. Some polarimetric parameters of the uterine cervix can be correlated with the gestational age. The uterine cervix's polarimetric analysis could make it possible to accurately predict the term of childbirth and be used as a screening tool for preterm birth.

DETAILED DESCRIPTION:
Interventional research protocol involving the human person relating to a medical device. This is a prospective, not randomized, monocentric study. Prematurity accounts for around 11% of births worldwide. In France, around 60,000 children (7.4%) are born each year prematurely. The term of gestation has a strong impact on mortality, severe neonatal morbidity, and child development. For this reason, premature birth represents a major public health issue. The means to reliably predict a premature birth are still ineffective. The medical device used in this research is a Mueller polarimetric colposcope which appears to be a powerful tool for evaluating the process of remodeling of cervical microstructure during pregnancy.

Mueller polarimetric imaging is the only technique that enables obtaining the comprehensive polarimetric characterization of a sample. Two groups are considered for this study: i) patients at low risk of premature birth (Group 1); ii) patients at high risk of premature birth (Group 2).

This study's main objective is to determine, for the two groups of patients, the best "polarimetric biomarkers" which make it possible to define an optimal "polarimetric score" reflecting the state of the cervical microstructure throughout its remodeling process during pregnancy.

This "Polarimetric Score" will be able to predict the term of childbirth and used as a screening tool for prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Major patient.
* Single pregnancy.
* Baseline ≥ 20 amenorrhea week for group 1 and baseline ≥ 20 amenorrhea week and <37 amenorrhea week for group 2.
* Dating obtained by ultrasound of the 1st trimester.
* Written and informed consent.

  * Group 1 (low risk):

Asymptomatic patient benefiting from usual follow-up in the maternity hospital.

> Group 2 (high risk): Symptomatic patient with cervical changes objectified by endovaginal ultrasound of the cervix with an effective length of <20mm.

Asymptomatic patient with a history of premature delivery or late miscarriage and cervical changes objectified by endovaginal ultrasound of the cervix with an effective length of <20mm."

Exclusion Criteria:

* Known uterine malformation or suspected uterine malformation.
* Pregnancy circled.
* Premature rupture of membranes.
* Suspicion of chorioamnionitis.
* Abundant active bleeding hindering the visualization of the cervix.
* History of conization.
* Imminent childbirth.
* Known medical indication at a birth <37 amenorrhea week (severe pre-eclampsia, severe intrauterine growth retardation, hemorrhagic placenta previa, fetal malformations,….).
* Examination of the cervix under speculum not possible.
* Lack of social coverage (AME).
* Limited understanding.
* Participation in another intervention research.

  > Group1 (Low risk):
* History of spontaneous premature labor.
* History of late miscarriage.
* History of premature rupture of membranes."

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Polarimetric parameters in population with a low-risk of premature birth | 6 months
  The principal outcome will be determining the best "polarimetric biomarkers" able to monitor and quantify the uterine cervix's modifications in a population with a low risk of premature birth. Specifically, the "polarimetric biomarkers" are the most relevant polarimetric parameters (or a combination of them) characterizing the cervical microstructure modifications during a normal pregnancy. They can be the main polarimetric parameters obtained from the measured Mueller matrices using different algebraic methods.
  One example of a polarimetric parameter that can be assessed is the Phase Retardance, measured in degrees at different wavelengths. It characterizes the anisotropy of the tissue.
Polarimetric biomarkers in population with a low-risk of premature birth | 6 months
  A polarimetric parameter that can be assessed is the azimuth of the Phase Retardance, measured in degrees at different wavelengths. It characterizes the orientations of the microscopic fibrous structures (such as the collagen) in the tissue.
Parameters Polarimetric in population with a low-risk of premature birth | 6 months
  A polarimetric parameter that can be assessed is the Depolarization, measured in arbitrary units at different wavelengths. It characterizes the scattering properties of the tissue.

SECONDARY OUTCOMES:
Polarimetric parameters in population with a high-risk of premature birth | 6 months
  A polarimetric parameter that can be assessed is the azimuth of the Phase Retardance, measured in degrees at different wavelengths. It characterizes the orientations of the microscopic fibrous structures (such as the collagen) in the tissue.
Polarimetric biomarkers in population with a high-risk of premature birth | 6 months
  A polarimetric parameter that can be assessed is the Depolarization, measured in arbitrary units at different wavelengths. It characterizes the scattering properties of the tissue.
Parameters polarimetric in population with a high-risk of premature birth | 6 months
  The principal outcome will be determining the best "polarimetric biomarkers" able to monitor and quantify the uterine cervix's modifications in a population with a high risk of premature birth. Specifically, the "polarimetric biomarkers" are the most relevant polarimetric parameters (or a combination of them) characterizing the cervical microstructure modifications during a normal pregnancy. They can be the main polarimetric parameters obtained from the measured Mueller matrices using different algebraic methods.
  One example of a polarimetric parameter that can be assessed is the Phase Retardance, measured in degrees at different wavelengths. It characterizes the anisotropy of the tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LUTON, Pr, Principal Investigator — Obstetrics gynecology department - Bicetre hospital, Kremlin Bicetre, France
Locations (1):
- Hospital Bicêtre - Gynecology-Obstetrics Department, Le Kremlin-Bicêtre, France, France